CLINICAL TRIAL: NCT05598294
Title: Can Wearable Technology Products Change Our Patient Management in Laparoscopic Colorectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Kamil Erozkan, Clinical Fellow, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AnkaraUSurgOnc
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Ambulation Difficulty; Physical Examination
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard treatment and mobilization recommendations will be given to this group.
- Mobilization Group (Experimental): Mobilization of patients will be encouraged.
  Interventions: Procedure: Mobilization recommendations

INTERVENTIONS:
Procedure: Mobilization recommendations — Standard mobilization recommendations will be given to all patients, and feedback will be given to the intervention group to increase the number of steps 4 times a day according to the daily targeted number of steps.
  Arms: Mobilization Group

SUMMARY:
The clinical progress of the patients whose mobilization the investigators follow up with wearable technology products will be observed in the early postoperative period until discharge. In this way, the investigators primarily aim to examine whether the bowel movements of our more mobilized patients return earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic abdominal surgery
* Colorectal cancer patients
* Curative surgeries
* Stage 0,1,2,3 patients

Exclusion Criteria:

* Patients who cannot walk
* Patients converted to open procedure
* Patients with ostomy
* Patients for whom laparoscopy is contraindicated
* Palliative surgeries
* Patients with distant organ metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to start flatus | 1 year

SECONDARY OUTCOMES:
Rate of Complications | 1 year
Length of stay | 1 year
Rate of Mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Faculty of Medicine, Surgical Oncology Department, Ankara
  - Ankara University, Ankara

IPD SHARING:
Plan to Share IPD: No
If requested, individual participant data (IPD) will be shared via e-mail after the reason has been evaluated.

REFERENCES:
- [Background] Daskivich TJ, Houman J, Lopez M, Luu M, Fleshner P, Zaghiyan K, Cunneen S, Burch M, Walsh C, Paiement G, Kremen T, Soukiasian H, Spitzer A, Jackson T, Kim HL, Li A, Spiegel B. Association of Wearable Activity Monitors With Assessment of Daily Ambulation and Length of Stay Among Patients Undergoing Major Surgery. JAMA Netw Open. 2019 Feb 1;2(2):e187673. doi: 10.1001/jamanetworkopen.2018.7673. PMID 30707226
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Heron N, Tully MA, McKinley MC, Cupples ME. Physical activity assessment in practice: a mixed methods study of GPPAQ use in primary care. BMC Fam Pract. 2014 Jan 15;15:11. doi: 10.1186/1471-2296-15-11. PMID 24422666
- [Result] Ganer Herman H, Kleiner I, Tairy D, Gonen N, Ben Zvi M, Kovo M, Bar J, Weiner E. Effect of Digital Step Counter Feedback on Mobility After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jun;135(6):1345-1352. doi: 10.1097/AOG.0000000000003879. PMID 32459426